CLINICAL TRIAL: NCT04696445
Title: Pharmacokinetics of Morphine and Oxycodone in Frail Elderly Undergoing Cardiac Surgery - AGE AWARE II
Brief Title: Pharmacokinetics of Morphine and Oxycodone in Frail Elderly Undergoing Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: St. Antonius Hospital (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, dr. P. Noordzij, Principal Investigator, St. Antonius Hospital
Other Study IDs: NL71713.100.20; 2020-001462-10 (EudraCT Number)
Record Dates: First submitted 2020-10-22; First posted 2021-01-06 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Opioid Use; Side Effect of Drug; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine; Oxycodone; Solutions; Injections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Morphine & Oxycodone — Morphine and Oxycodone are used in daily practice as part of standard care. Morphine and Oxycodone will be acquired through the clinical pharmacy of St Antonius and administered according to the standard postoperative pain protocol.
  Other Names: Morphine HCl CF 10mg/mL solution for injection / infusion; OxycodoneHCl G.L. tablet 5/10mg.; OxycodoneHCl Retard Lannacher 5/10/20 mg.

SUMMARY:
* Single centre observational cohort study.
* 20 older patients undergoing cardiac surgery who receive standard of care pain treatment.
* Postoperative ICU: blood sampling to determine morphine and metabolite (M3G, M6G, noroxycodone and oxymorphone) pharmacokinetics
* After ICU discharge on general ward: blood sampling to determine morphine, oxycodone and metabolite (M3G, M6G, noroxycodone and oxymorphone) pharmacokinetics
* During study monitoring of pain scores, total opioid consumption, side effects (e.g. nausea, vomiting, pruritus), sedation and delirium scores.

DETAILED DESCRIPTION:
Postoperative pain after cardiac surgery in elderly patients is common and leads to postoperative complications. Opioids play an important role in treatment of postoperative pain after cardiac surgery. In frail elderly after cardiac surgery however dosing schemes for opioids are still unknown, potentially leading to inadequate treatment of pain and/or safety issues.

* Single center observational cohort study
* The study population includes frail patients ≥70 years undergoing elective cardiac surgery.
* Primary endpoints of this study is the concentration of morphine, oxycodone and metabolites in blood over time on behalf of pharmacokinetic modelling.
* Secondary endpoints of this study are the pharmacodynamic parameters of morphine, oxycodone and metabolites (M3G, M6G, noroxycodone and oxymorphone) in blood in frail patients; such as pain scores, postoperative opioid consumption, vital signs, side effects of opioids and the influence of covariates such as frailty, serum creatinine, Glomerular Filtration Rate (GFR) on the pharmacokinetics and pharmacodynamics of morphine and oxycodone.

ELIGIBILITY:
Inclusion Criteria:

* ≥70 years undergoing elective cardiac surgery.

Exclusion Criteria:

* Patients undergoing transcatheter aortic valve replacement or mitral valve repair
* Contra-indication for morphine and/or oxycodone

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population includes 20 patients ≥70 years undergoing elective cardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-11-26 (Actual); Study Completion 2021-11-26 (Actual)

PRIMARY OUTCOMES:
M3G concentration in blood over time | Until three consecutive days after ICU discharge
  Analysis of serum concentrations of M3G, metabolite of morphine, for pharmacokinetic modelling
M6G concentration in blood over time | Until three consecutive days after ICU discharge
  Analysis of serum concentrations of M6G, metabolite of morphine, for pharmacokinetic modelling
Noroxycodone concentration in blood over time | Until three consecutive days after ICU discharge
  Analysis of serum concentrations of Noroxycodone, metabolite of oxycodone, for pharmacokinetic modelling
Oxymorphone concentration in blood over time | Until three consecutive days after ICU discharge
  Analysis of serum concentrations of Oxymorphone, metabolite of oxycodone, for pharmacokinetic modelling

SECONDARY OUTCOMES:
Numeric Rating Scale (NRS; 0-10, 0 = none, 10 = severe) | Until three consecutive days after ICU discharge
  NRS as pain measurement scale, reported by nurse in standard care, for pharmacodynamic modelling
Postoperative opioid consumption | Until three consecutive days after ICU discharge
  Postoperative opioid consumption, mg per 24 hour, for pharmacodynamic modelling
Side effects of opioids | Until three consecutive days after ICU discharge
  Side effects of opioids (pruritis, vomiting, constipation, nausea), dichotomous (yes/no) each day by nurse/researcher, for pharmacodynamic modelling
Vital sign observation: bloodpressure (in mmHg) by nurse | Until three consecutive days after ICU discharge
  Systolic and diastolic bloodpressure (SBP, DBP), reported by nurse in standard care for pharmacodynamic modelling
Vital sign observation: heartrate (in beats/minute) by nurse | Until three consecutive days after ICU discharge
  Heartrate (HR) reported by nurse in standard care for pharmacodynamic modelling
Vital sign observation: saturation (in %) by nurse | Until three consecutive days after ICU discharge
  Saturation (SpO2), reported by nurse in standard care for pharmacodynamic modelling

CONTACTS AND LOCATIONS:
Locations (1):
- St Antonius hospital, Nieuwegein, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Plan to Share IPD: Undecided